CLINICAL TRIAL: NCT06203067
Title: Type 1 Together: A Peer Mentorship Program to Bolster Use of Continuous Glucose Monitoring Systems Among Adolescents With Type 1 Diabetes
Brief Title: Type 1 Together: A Peer Mentorship Program to Bolster Use of CGM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Paul Enlow, Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1990806; P20GM144270 (NIH); 5438 (Other: NIGMS Sub-Project ID)
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 Together (Experimental): In Type 1 Together, families will work with other families who have experience using CGM (Peer Mentors) to overcome common barriers to CGM use. Families in the Type 1 Together program will also have access to CGM-specific educational materials, a digital journal to facilitate patient-provider communication around issues with CGM, and social determinant of health screening and intervention with a diabetes community health worker.
  Interventions: Behavioral: Type 1 Together
- Standard of Care (Active Comparator): Quarterly clinic visits with endocrinology provider.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Standard of Care — Quarterly clinic visits with endocrinology provider.
  Arms: Standard of Care
Behavioral: Type 1 Together — In Type 1 Together, families will work with other families who have experience using CGM (Peer Mentors) to overcome common barriers to CGM use. Families in the Type 1 Together program will also have access to CGM-specific educational materials, a digital journal to facilitate patient-provider communication around issues with CGM, and social determinant of health screening and intervention with a diabetes community health worker.
  Arms: Type 1 Together

SUMMARY:
The goal of this clinical trial is to evaluate a new way of helping adolescents with type 1 diabetes consistently use continuous glucose monitoring systems (CGM).

Families who participate will be assigned by chance to one of two groups. One group will continue to see their Endocrinology provider who can give recommendations on ways to use CGM.

The other group will be in our Type 1 Together program for 6 months. This will include:

1. Monthly meetings with a community health worker with expertise in type 1 diabetes self-management,
2. Access to CGM-specific educational resources hosted on a mobile app, and
3. Meeting at least monthly with a mentor family who will provide mentorship on using CGM consistently.

The main questions the study aims to answer are:

1. Do families like the Type 1 Together program?
2. Do more families in the Type 1 Together program have better attitudes towards CGM, use CGM more consistently, and have lower HbA1c?
3. Does the Type 1 Together program reduce racial and ethnic differences in attitudes towards CGM, consistent use of CGM, and HbA1c?

ELIGIBILITY:
Inclusion Criteria:

* 12 to 17 years old
* Diagnosed with type 1 diabetes for at least 6 months
* Does not use CGM OR uses CGM < 24 out of the past 30 days
* Use CGM 24 to 30 of the past 30 days but most recent HbA1c was 9% or more
* Able to read and write in English

Exclusion Criteria:

* Type 1 diabetes due to other medical condition (e.g., cystic fibrosis)
* Intellectual disability
* Severe psychiatric comorbidities

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | 6 months post-enrollment
  How acceptable youth and caregivers find Type 1 Together. This information will be collected only from participants in the experimental arm using the Acceptability of Intervention Measure (scores range 1-5 with higher scores indicating greater acceptability).
Perceptions of continuous glucose monitoring systems | Baseline and 3, 6, 9, and 12 months post-enrollment.
  Youth perceptions of the benefits and burdens of using continuous glucose monitoring systems will be assessed using the CGM Benefits and Burdens Scales (scores range 1-5 with higher scores indicating greater perceived benefits or burdens).
Continuous Glucose Monitoring System Use | Baseline and 3, 6, 9, and 12 months post-enrollment
  The number of days a patient wore their continuous glucose monitoring system at least 12 hours over the past month.
HbA1c | Baseline and 3, 6, 9, and 12 months post-enrollment
  HbA1c expressed as a percentage of glycosylated hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Hospital, Delaware, Wilmington, Delaware, United States